CLINICAL TRIAL: NCT07332247
Title: An Open-Label, Randomized Controlled Phase II Clinical Trial of PD-1 Inhibitor Plus Chemotherapy Followed by Immediate Versus Selective Re-irradiation for Locally Advanced Recurrent Nasopharyngeal Carcinoma
Brief Title: PD-1 Inhibitor Plus Chemotherapy Followed by Immediate Versus Selective Re-irradiation for Locally Advanced Recurrent NPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-205
Record Dates: First submitted 2025-12-24; First posted 2026-01-12 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Nasopharangeal Cancer; Recurrent Nasopharynx Carcinoma
Keywords: Locally Advanced Recurrent Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective re-irradiation group (Other): PD-1 inhibitor maintenance + Selective re-irradiation:
  PD-1 inhibitor maintenance therapy:Toripalimab 240 mg IV on day 1 every 3 weeks, or Tislelizumab 200 mg IV on day 1 every 3 weeks, or Camrelizumab 200 mg IV on day 1 every 3 weeks, continued until disease progression (per RECIST v1.1; if progression occurs in the nasopharynx or neck, re-irradiation will be administered and PD-1 maintenance will continue until subsequent progression), unacceptable toxicity, patient withdrawal, or a maximum treatment duration of 2 years.
  Interventions: Radiation: Selective re-irradiation
- Immediate re-irradiation group (Other): Immediate re-irradiation + PD-1 inhibitor Maintenance:
  Re-irradiation will be administered Immediately. PD-1 inhibitor maintenance therapy: Toripalimab 240 mg IV on day 1 every 3 weeks, or Tislelizumab 200 mg IV on day 1 every 3 weeks, or Camrelizumab 200 mg IV on day 1 every 3 weeks, continued until disease progression (per RECIST v1.1), unacceptable toxicity, patient withdrawal, or a maximum treatment duration of 2 years.
  Interventions: Radiation: Immediate re-irradiation

INTERVENTIONS:
Radiation: Selective re-irradiation — PD-1 inhibitor maintenance + Selective re-irradiation PD-1 inhibitor maintenance therapy:Toripalimab 240 mg IV on day 1 every 3 weeks, or Tislelizumab 200 mg IV on day 1 every 3 weeks, or Camrelizumab 200 mg IV on day 1 every 3 weeks, continued until disease progression (per RECIST v1.1; if progression occurs in the nasopharynx or neck, re-irradiation will be administered and PD-1 maintenance will continue until subsequent progression), unacceptable toxicity, patient withdrawal, or a maximum treatment duration of 2 years.
  Arms: Selective re-irradiation group
Radiation: Immediate re-irradiation — Immediate re-irradiation + PD-1 inhibitor Maintenance:
  Re-irradiation will be administered Immediately. PD-1 inhibitor maintenance therapy: Toripalimab 240 mg IV on day 1 every 3 weeks, or Tislelizumab 200 mg IV on day 1 every 3 weeks, or Camrelizumab 200 mg IV on day 1 every 3 weeks, continued until disease progression (per RECIST v1.1), unacceptable toxicity, patient withdrawal, or a maximum treatment duration of 2 years.
  Arms: Immediate re-irradiation group

SUMMARY:
This phase II randomized trial evaluates PD-1 inhibitor plus chemotherapy followed by immediate versus selective re-irradiation in locally advanced recurrent nasopharyngeal carcinoma. The study aims to determine whether sequential radiotherapy provides additional survival benefit beyond systemic immunochemotherapy.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is prevalent in Southern China, and 10~15% of patients experience local recurrence, which presents significant treatment challenges. PD-1 inhibitor plus gemcitabine-cisplatin (GP) has become the standard first-line therapy for recurrent/metastatic NPC. However, the survival benefit of adding sequential re-irradiation after GP + PD-1 in locally advanced recurrent nasopharyngeal carcinoma remains uncertain.This phase II randomized trial aims to compare immediate versus selective re-irradiation following PD-1 inhibitor plus GP in locally advanced recurrent NPC, to determine whether sequential re-irradiation provides additional survival benefit without excessive toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years, any gender.
2. Local recurrence (with or without regional recurrence) more than one year after radical treatment and unsuitable for surgery.
3. Pathologically confirmed non-keratinizing nasopharyngeal carcinoma (WHO type II or III).
4. Achieved complete response (CR) or partial response (PR) after 4-6 cycles of chemotherapy plus PD-1 inhibitor therapy.
5. ECOG performance status 0-1.
6. Expected survival ≥ 3 months.
7. No prior radiotherapy, chemotherapy, immunotherapy, or biological therapy for recurrent nasopharyngeal carcinoma
8. No contraindications to immunotherapy, chemotherapy, or re-irradiation.
9. Adequate organ function within 14 days before first dose, defined as:

   Hematology：Hemoglobin ≥ 90 g/L，ANC ≥ 1.5 × 10⁹/L，Platelet count ≥ 100 × 10⁹/L Renal Function：Creatinine ≤ 1.5 × ULN, or creatinine clearance (CrCl) / eGFR ≥ 60 mL/min Liver Function：Total bilirubin ≤ 1.5 × ULN，AST and ALT ≤ 2.5 × ULN, or ≤ 5 × ULN in the presence of liver metastases
10. INR or PT ≤ 1.5 × ULN, unless on therapeutic anticoagulation and values within therapeutic range，APTT ≤ 1.5 × ULN, unless on therapeutic anticoagulation and values within therapeutic range.

Exclusion Criteria:

1. Presence of grade 3 or higher late radiation toxicity (excluding skin, subcutaneous tissue, and mucosa) at the time of recurrence
2. Prior anti-tumor therapy for recurrent nasopharyngeal carcinoma, including radiotherapy, chemotherapy, surgery, or immunotherapy.
3. Prior treatment with PD-1/PD-L1 or CTLA-4 inhibitors.
4. History of other malignancies within the past 5 years, except adequately treated basal cell carcinoma, squamous cell skin cancer, or in-situ cervical cancer.
5. Active autoimmune disease or history of autoimmune disease requiring systemic treatment (e.g., corticosteroids, immunosuppressants) within the past 2 years, except for stable hypothyroidism, type 1 diabetes mellitus, or resolved childhood asthma/atopy.
6. Known history of active pulmonary tuberculosis (TB). Suspected active TB must be excluded by chest X-ray, sputum examination, and assessment of clinical signs and symptoms.
7. Hepatitis B: HBsAg positive with peripheral blood HBV DNA ≥ 1000 copies/mL
8. Hepatitis C: HCV antibody positive, eligible only if HCV RNA is negative
9. HIV infection
10. Clinically significant cardiovascular disease (e.g., uncontrolled hypertension, unstable angina, myocardial infarction within 6 months, congestive heart failure ≥ NYHA class II, or serious arrhythmia).
11. Interstitial lung disease, non-infectious pneumonitis, or history of ≥ grade 2 pneumonitis.
12. Major surgery within 4 weeks before enrollment, or unhealed surgical wound.
13. Pregnant or breastfeeding women, or those planning pregnancy during the study period.
14. Known allergy or hypersensitivity to study drugs or their excipients.
15. Any condition that, in the investigator's judgment, would interfere with trial participation or interpretation of results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2026-02-03 (Estimated); Primary Completion 2032-02-03 (Estimated); Study Completion 2035-02-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 year
  the time from the date of randomization to the date of death due to any cause.

SECONDARY OUTCOMES:
Progression free-survival | 3 year
  the time from randomization to the first objectively documented disease progression, or death from any cause, whichever occurs first.
Progression free-survival 2 | 3 year
  the time from randomization to second/subsequent disease progression after initiation of new anticancer therapy, or death from any cause, whichever occurs first
Locoregional progression-free survival | 3 year
  the time from random assignment to the occurrence of a locoregional progression.
Distant progression-free survival | 3 year
  Defined as the time from random assignment to the occurrence of a distant progression.
Incidence of Acute and Late Toxicity | 3 year
  Incidence of acute toxicity is calculated for each adverse event respectively and severity is evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE) 5.0 criteria. Late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme.
Quality of life (QoL) | 3 year
  Assessed using the EORTC QLQ-C30 (v3.0)
Quality of life (QoL) | 3 year
  Assessed using the EORTC QLQ-H&N35 (v1.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No